CLINICAL TRIAL: NCT01876069
Title: Comparing Newly Developed PreCore Needle With Conventional Fine Needle in Endoscopic Ultrasonography-guided Sampling of Suspected Unresectable Pancreatic Cancer
Brief Title: Comparing Newly Developed PreCore Needle With Conventional Fine Needle in Suspected Unresectable Pancreatic Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: Olympus (Industry)
Responsible Party: Principal Investigator, Kwang Hyuck Lee, Assistant Professor, Samsung Medical Center
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-02-018
Record Dates: First submitted 2013-06-04; First posted 2013-06-12 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 22 gauge ProCore needle aspiration (Active Comparator): EUS-guided pancreatic mass aspiration with 22 gauge ProCore needle
  Interventions: Device: 22 gauge ProCore needle aspiration
- 22 gauge Fine needle aspiration (Active Comparator): EUS-guided pancreatic mass aspiration with 22 gauge Fine needle
  Interventions: Device: 22 gauge Fine needle aspiration

INTERVENTIONS:
Device: 22 gauge ProCore needle aspiration — Pancreatic mass evaluation through the 22 gauge ProCore needle aspiration
  Other Names: EchoTip® ProCore™ High Definition Ultrasound Biopsy Needle
  Arms: 22 gauge ProCore needle aspiration
Device: 22 gauge Fine needle aspiration — Pancreatic mass evaluation through the 22 gauge Fine needle aspiration
  Other Names: 22 gauge, EN-SHOT2 Side Port Aspiration Needle
  Arms: 22 gauge Fine needle aspiration

SUMMARY:
Background:

Pancreatic cancer is associated with a poor prognosis. Therefore, rapid and accurate diagnosis of a pancreatic mass is important to direct patient management. Endoscopic ultrasonography-guided fine needle aspiration (EUS-FNA) is the current standard for sampling pancreatic mass lesions, with diagnostic accuracy of 78% to 95%. But, the EUS-FNA has some limitations include stromal cell tumors and lymphomas may be difficult to diagnose. To overcome these limitations, a new needle device with ProCore reverse-bevel technology was developed recently.

Aims:

The objective of this prospective study is to compare the rate of diagnostic sufficiency in the EUS sampling by using newly developed ProCore needle with conventional FNA needle in suspected unresectable pancreatic cancer. We will also compare the safety, the yield of histologic core tissue and the cost-effectiveness between these modalities.

DETAILED DESCRIPTION:
Patient:

Newly diagnosed pancreatic cancer patient whose cancer lesion is suspected unresectable in diagnostic imaging such as CT or MRI

Procedure:

Each EUS-guided FNA and ProCore aspiration will performed twice in same patient. The priority of order will be given by randomization assignment.

The number of patients required:

Total sixty five patients will be required.

ELIGIBILITY:
Inclusion Criteria:

* Patients who agree to participate in research
* 18 years of age and older patients less than 80 years old
* Patients who have suspected unresectable pancreatic cancer in imaging studies

Exclusion Criteria:

* Contraindication to endoscopy
* Patients younger than 18 years old or older than 80 years old
* Bleeding tendency
* Cardiopulmonary dysfunction
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2013-07; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The rates of diagnostic sufficiency | Up to 1 year
  The rates of diagnostic sufficency will be assessed by the pathologist as the proportion of definate diagnosis from cytology and histology within 2 passes of each procendure

SECONDARY OUTCOMES:
The presence of histologic core | Up to 1 year
  The presence histologic core means the gain of tissue, not clustered cells, through each procedure. It will be also assessed by the pathologist.

OTHER OUTCOMES:
Procedure related complications | Up to 1 year
  Investigate the occurrence of complications such as bleeding, perforation, pancreatitis, infection. Not only complications, but the size and location of lesion, puncture routes will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Kwang Hyuck Lee, MD., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea